CLINICAL TRIAL: NCT04225416
Title: The ePISTLE Study: Perceptions of Illness Severity, Treatment Goals and Life Expectancy
Brief Title: Perceptions of Illness Severity, Treatment Goals and Life Expectancy
Acronym: ePISTLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 18HH4336
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Hemodialysis; Peritoneal Dialysis
Keywords: hemodialysis; peritoneal dialysis
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemodialysis patients: Patients undergoing hemodialysis
  Interventions: Other: Questionnaire/Structured Interview
- Peritoneal dialysis patients: Patients undergoing peritoneal dialysis
  Interventions: Other: Questionnaire/Structured Interview

INTERVENTIONS:
Other: Questionnaire/Structured Interview — No intervention

SUMMARY:
This study is exploring symptom burden, health experiences and expectations of treatment and survival of seriously ill dialysis patients and their physicians.

DETAILED DESCRIPTION:
Sharing and communicating information with patients is an integral part of medical care, yet research has shown that disparities exist between physicians and patient perceptions of illness severity. In renal medicine, along with many other specialties, expected prognosis can affect treatment offered.Thus appreciating and understanding one's prognosis can influence patients and relatives' expectations for treatment and guide discussions regarding quality of life.

Previous work has highlighted disparities in the United States between expectations of survival of seriously ill haemodialysis patients and their physicians. The investigators plan to repeat this study within the United Kingdom, to see whether similar issues occur and to elucidate current practice on discussions of prognosis, symptom burden and transplant candidacy. The investigators hope to identify where care can be improved and to enable patients to better make informed decisions on treatment and goals of care.

Part one of the study is to repeat this study in haemodialysis patients in the United Kingdom. This has been completed and published (2021) at https://www.kireports.org/article/S2468-0249(21)00103-0/fulltext.

Part two of the study is to extend the study to peritoneal dialysis patients in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Haemodialysis patients 18-100 years old, with a predicted mortality risk of >20% in the next year, their close person and staff members (nurse and doctor) caring for the patient.
* Peritoneal dialysis patients 18-100 years old, with a predicted mortality risk of >20% in the next year, their close person and staff members (nurse and doctor) caring for the patient.

Exclusion Criteria:

* Patients on home haemodialysis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Current practice regarding discussion of prognosis with seriously ill dialysis patients, to better understand the dissonance between physician and patient beliefs on prognosis, transplant candidacy and goals of care. | Through study completion, an average of 2 years
  Completion of questionnaire or structured interview

SECONDARY OUTCOMES:
Number of dialysis patients who are more optimistic about prognosis and transplant candidacy than their nephrologists | Through study completion, an average of 2 years
  Completion of questionnaire or structured interview
Patients' prognostic expectations are associated with their treatment preferences | Through study completion, an average of 2 years
  Completion of questionnaire or structured interview
Number of patients with dialysis associated symptoms as assessed by IPOS Renal (https://pos-pal.org/maix/ipos-renal-in-english.php). | 7 days
  Completion of questionnaire or structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Edwina Brown, MBChB, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided